CLINICAL TRIAL: NCT00446680
Title: Long Term Administration of Inhaled Dry Powder Mannitol In Cystic Fibrosis - A Safety and Efficacy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Brett Charlton, Pharmaxis Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPM-CF-301
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Cystic Fibrosis
Keywords: Mannitol; Cystic Fibrosis; Mucolytic; Exacerbation; FEV1; Quality of Life
MeSH Terms: conditions — Cystic Fibrosis | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Mannitol
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mannitol — 400mg BD for 6 months followed by a 6 month open label period
  Arms: 1
Drug: placebo — placebo BD for 6 months
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy and safety of chronic treatment with inhaled dry powder mannitol in subjects with cystic fibrosis. Previous studies have demonstrated an improvement in lung function related to small airways obstruction and a significant improvement in respiratory symptoms and quality of life after a 2 week treatment with mannitol. This current study seeks to support these early findings and to extend the evidence to support its use as a mucoactive therapy in cystic fibrosis. In particular, the hypothesis that enhanced mucus clearance will improve the lung function and clinical presentation in this population, will be investigated. We also hypothesize that enhanced mucociliary clearance will result in a sustained reduction in mucus load, thus providing less opportunity for bacteria to proliferate, affording a reduction in antibiotic use and hospitalizations. The initial 6 month blinded phase will be followed with an additional 6 months of open label treatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Confirmed diagnosis of cystic fibrosis
* Aged > 6 years
* FEV1 >30 % and < 90% predicted
* Able to perform all the techniques necessary to measure lung function

Main Exclusion Criteria:

* "Terminally ill" or listed for lung transplantation
* Had a lung transplant
* Using nebulised hypertonic saline
* Significant episode of haemoptysis (>60 mL) in the three months prior to enrolment
* Recent myocardial infarction or cerebral vascular accident
* Breast feeding or pregnant, or plan to become pregnant while in the study participating in another investigative drug study, parallel to, or within 4 weeks of study entry
* Allergy or intolerance to mannitol
* Using beta blockers
* Have a condition or be in a situation which in the Investigator's opinion may put the subject at significant risk, may confound results or may interfere significantly with the patient's participation in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the effects of 400 mg twice-daily administration of IDPM on FEV1 in patients with CF compared to control | 6 months

SECONDARY OUTCOMES:
To determine the effects of 400 mg twice-daily administration of IDPM on FEV1 in patients with CF on existing RhDNase treatment compared to control. (key objective) | 6 months
Reduces pulmonary exacerbations in those taking RhDNase as a sub-group and in the total cohort (key objective) | 6 months / 12 months
Improves quality of life (key objective) | 6 months
Reduces days on IV antibiotics, rescue oral or inhaled antibiotics | 6 months / 12 months
Reduces days in hospital due to pulmonary exacerbations | 6 months / 12 months
Improves other measures of lung function | 6 months
Demonstrates an appropriate safety profile (adverse events, haematology, biochemistry, change in bronchodilator response, sputum microbiology, physical examination) | 6 months / 12 months
Reduces hospital and community care costs | 6 months / 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brett Charlton, MBBS, Study Director — Pharmaxis Ltd Australia; Dr Diana Bilton, Principal Investigator — Papworth Hospital NHS Foundation Trust; Dr Philip Robinson, Principal Investigator — Royal Children's Hospital
Locations (29):
- Australia (6):
  - Childrens Hospital at Westmead, Sydney, New South Wales
  - Sydney Childrens Hospital, Sydney, New South Wales
  - Royal Brisbane Children's Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Childrens Hospital, Melbourne, Victoria
- Ireland (4):
  - Beaumont Hospital, Dublin
  - National Children's Hospital, Dublin
  - Our Lady's Hospital for Sick Children, Dublin
  - St Vincent's University Hospital, Dublin
- United Kingdom (19):
  - Alder Hey Children's Hospital, West Derby, Liverpool
  - Belfast City Hospital, Belfast, Northern Ireland
  - Children's Hospital for Wales, Cardiff, Wales
  - Llandough Hospital, Cardiff, Wales
  - Birmingham Children's Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Bristol Royal Infirmary, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Papworth Hospital, Cambridge
  - Seacroft Hospital, Leeds
  - Cardiothoracic Centre, Liverpool
  - The London Chest Hospital, London
  - Freeman Hospital, Newcastle
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Northern General Hospital, Sheffield
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Yang C, Montgomery M. Dornase alfa for cystic fibrosis. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD001127. doi: 10.1002/14651858.CD001127.pub5. PMID 33735508
- [Derived] Nevitt SJ, Thornton J, Murray CS, Dwyer T. Inhaled mannitol for cystic fibrosis. Cochrane Database Syst Rev. 2020 May 1;5(5):CD008649. doi: 10.1002/14651858.CD008649.pub4. PMID 32358807
- [Derived] Bilton D, Robinson P, Cooper P, Gallagher CG, Kolbe J, Fox H, Jaques A, Charlton B; CF301 Study Investigators. Inhaled dry powder mannitol in cystic fibrosis: an efficacy and safety study. Eur Respir J. 2011 Nov;38(5):1071-80. doi: 10.1183/09031936.00187510. Epub 2011 Apr 8. PMID 21478216